CLINICAL TRIAL: NCT05076045
Title: Immediate Effects of Personal Sound Amplification Products on Speech Processing
Brief Title: Effects of PSAPs on Speech Processing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rotman Research Institute at Baycrest (Other)
Responsible Party: Principal Investigator, Claude Alain, Senior Scientist, Rotman Research Institute at Baycrest
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PSAPs2021
Record Dates: First submitted 2021-09-20; First posted 2021-10-13 (Actual); Results first posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Hearing Loss, Age-Related
Keywords: Hearing loss; Speech processing; Speech-in-noise; Aging
MeSH Terms: conditions — Presbycusis; Hearing Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personal sound amplification products (Experimental): Speech perception will be evaluated using personal sound amplification products.
  Interventions: Device: Personal sound amplification products
- Control (No Intervention): Speech perception will be evaluated without using hearing devices.

INTERVENTIONS:
Device: Personal sound amplification products — Participants will be tested with bilateral personal sound amplification products.
  Arms: Personal sound amplification products

SUMMARY:
Mild to moderate hearing loss remains undertreated, largely because of the high cost of hearing aids. A promising and much less expensive alternative is the use of personal sound amplification products (PSAPs), which are electronic, portable, over-the-counter devices that amplify sound. Studies have shown that the use of PSAPs provides significant hearing benefits and improves the quality of life for older adults with mild to moderate hearing loss. However, there is insufficient data to determine the impact of PSAPs use on speech processing in the brain.

The purpose of this study is to use electroencephalography (EEG) measurements to assess the neurobiological and behavioral effects of PSAPs on speech perception in noise in individuals with mild to moderate hearing loss.

The investigators expect that the PSAPs use will result in an immediate improvement in the ability to perceive speech-in-noise, supporting that these hearing devices may be a means of restoring communication skills in people with mild to moderate hearing loss. Behavioral benefits will be associated with increased brain activity in auditory regions and connectivity between auditory and speech regions in the brain.

DETAILED DESCRIPTION:
This study will consist of two sessions of 3 hours each. On one session, participants will perform the speech-in-noise task without hearing devices and on the other session, participants will perform the speech-in-noise task while wearing personal sound amplification products. The order of the sessions will be counterbalanced across participants. The speech-in-noise task consists in a word discrimination task in babble noise at three signal-to-noise ratios. On each trial, the task is to determine whether two words are identical or different.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed

Exclusion Criteria:

* Mother tongue not English
* Language impairment
* Dementia
* Cerebrovascular diseases
* Untreated vision impairment;
* Tinnitus and otologic disorders
* Cochlear implant
* History of prior hearing aid use
* Diagnosed addiction (alcohol or drugs)
* Significant medical or neurocognitive conditions or interventions likely to significantly impact cognitive function (e.g., epilepsy, stroke, traumatic brain injury with loss of consciousness > 5 minutes, brain tumor, multiple sclerosis, hepatitis C, developmental delay, electroconvulsive therapy)
* a diagnosis (based on the Diagnostic and Statistical Manual of Mental Disorders (DSM-5)) of major depressive disorder with active symptoms within 90 days of study entry, past or present psychosis, or other psychiatric disorders such as obsessive-compulsive disorder, generalized anxiety disorder, and bipolar disorder

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claude Alain, PhD, Principal Investigator — Rotman Research Institute at Baycrest Centre
Locations (1):
- Rotman Research Institute at Baycrest Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Demographic and health information, behavioral results, and EEG recordings will be shared on an open platform only if participants consent. The data will be anonymized using a random generic code. No personally identifiable data will be shared. The code and stimuli of the task will also be shared on the platform.
Supporting Information: Study Protocol, Analytic Code
Time Frame: The data will be shared when the article is published and will remain accessible as long as possible.
Access Criteria: Data will be shared on an open platform to be determined. The web address of the data sharing will be inserted in the article, and anyone can access the data from this link.

REFERENCES:
- [Derived] Perron M, Dimitrijevic A, Alain C. Rapid Brain Adaptation to Hearing Amplification: A Randomized Crossover Trial of Personal Sound Amplification Products. Trends Hear. 2025 Jan-Dec;29:23312165251375891. doi: 10.1177/23312165251375891. Epub 2025 Sep 5. PMID 40910451
- [Derived] Perron M, Lau B, Alain C. Interindividual variability in the benefits of personal sound amplification products on speech perception in noise: A randomized cross-over clinical trial. PLoS One. 2023 Jul 19;18(7):e0288434. doi: 10.1371/journal.pone.0288434. eCollection 2023. PMID 37467243

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 72 participants were screened for eligibility between March 1, 2022 and September 31, 2022 by telephone interview at Baycrest Hospital in Toronto, Canada.
Pre-assignment Details: 32 of the 72 participants were randomized. Of those who were not randomized, 22 did not meet the inclusion criteria, 14 declined to participate and four had other reasons.
Groups:
- Personal Sound Amplification Products First, Then Control: Participants were tested for speech-in-noise perception while using bilateral personal sound amplification products during the first session. After a one-week washout period, they were retested for speech-in-noise perception while not using a device.
- Control First, Then Personal Sound Amplification Products: Participants were tested for speech perception in noise while using no devices during the first session. After a one-week washout period, they were retested for speech-in-noise perception while using bilateral personal sound amplification products.
Period: First Intervention (3 Hours)
Arm/Group | Personal Sound Amplification Products First, Then Control | Control First, Then Personal Sound Amplification Products
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0
Period: Washout (1 Week)
Arm/Group | Personal Sound Amplification Products First, Then Control | Control First, Then Personal Sound Amplification Products
Started | 16 | 16
Completed | 15 | 13
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 3
Period: Second Intervention (3 Hours)
Arm/Group | Personal Sound Amplification Products First, Then Control | Control First, Then Personal Sound Amplification Products
Started | 15 | 13
Completed | 15 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Personal Sound Amplification Products First, Then Control | Control First, Then Personal Sound Amplification Products | Total
Number analyzed (Participants) | 15 | 13 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 74 (6.6) | 72.23 (6.25) | 73.18 (6.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 6 | 3 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 15 | 13 | 28

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Correct Responses With and Without PSAPs
Description: Percentage (%) of correct responses in the speech-in-noise task when using PSAPs and when using no device.
Time Frame: 1 hour
Population: All participants who completed all study visits were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: percentage of correct answers
Groups:
- Personal Sound Amplification Products: Participants were tested for speech-in-noise perception while using bilateral personal sound amplification products.
- Control: Participants were tested for speech perception in noise while using no devices.
Arm/Group | Personal Sound Amplification Products | Control
Number analyzed (Participants) | 28 | 28
percentage of correct answers | 85.2 [83.2 to 87.4] | 84.0 [81.9 to 86.0]
Statistical Analysis 1: Comparison: Personal Sound Amplification Products vs Control; Null hypothesis is that there was no difference in percentage of correct answers between PSAPs and Control. Data were analyzed using a linear mixed-effects (LME) model. The model included session (PSAPs, Control) and signal-to-noise ratio (SNR) as within-subject factors. Participants were included as a random factor; Test type: Superiority; p = 0.03, Mixed Models Analysis — This p-value has been adjusted using the Bonferroni correction. The threshold for statistical significance was p = 0.05 (two-sided); Results of the pairwise comparisons for the SNR by Session interaction in the linear mixed model analysis

2. Primary Outcome: Reaction Time With and Without PSAPs
Description: Reaction time (in milliseconds) in the speech-in-noise task when using PSAPs and when using no device.
Time Frame: 1 hour
Population: All participants who completed all study visits were included in the analysis. Data from one participant was lost due to a technical issue. Additionally, one participant was excluded because their reaction time values exceeded 3 times the interquartile range.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Personal Sound Amplification Products | Control
Number analyzed (Participants) | 26 | 26
milliseconds | 528.7 (155.1) | 502.0 (145.9)
Statistical Analysis 1: Comparison: Personal Sound Amplification Products vs Control; Null hypothesis is that there was no difference in reaction time between PSAPs and Control. Data were analyzed using a linear mixed-effects (LME) model. The model included session (PSAPs, Control) and signal-to-noise ratio as within-subject factors. Participants were included as a random factor; Test type: Superiority; p = 0.28, Mixed Models Analysis — The threshold for statistical significance was p = 0.05 (two-sided)

3. Primary Outcome: Quick Speech In Noise Score With and Without PSAPs
Description: Performance on the QuickSIN when using PSAPs and when using no device. The QuickSIN measures the signal-to-noise ratio loss. A high score indicates poorer speech understanding in noise.
Time Frame: 1 hour
Population: All participants who completed all study visits were included in the analysis.
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Personal Sound Amplification Products | Control
Number analyzed (Participants) | 28 | 28
dB | 3.6 (2.2) | 4.6 (2.4)
Statistical Analysis 1: Comparison: Personal Sound Amplification Products vs Control; Null hypothesis is that there was no difference in Quick Speech In Noise score between PSAPs and Control. The performance of the QuickSIN for the two sessions (PSAPs, Control) was compared using the Wilcoxon signed rank test on paired samples; Test type: Superiority; p = 0.005, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p = 0.05 (two-sided)

4. Primary Outcome: Alpha Power (8-12 Hz) During the Processing of the First Word in a Low Noise Condition, With and Without PSAPs
Description: Alpha power (8-12 Hz) for a cluster of temporoparietal electrodes (T7, TP7, CP5), measured between 50 and 500 ms after the onset of the first word of the speech-in-noise task, under a low noise condition (signal-to-noise ratio of +3 dB), with and without PSAPs. Alpha power was measured using temporal spectral evolution analysis with EEG. Values are baseline corrected with the pre-stimulus interval period (-500, 0 ms). Higher values indicate greater alpha power compared to the pre-stimulus interval period (i.e., event-related synchronization).
Time Frame: 1 hour
Population: One participant did not complete the EEG portion of the study. Two other participants were excluded due to noisy data.
Measure: Mean (Standard Deviation); unit: percentage of power change
Arm/Group | Personal Sound Amplification Products | Control
Number analyzed (Participants) | 25 | 25
percentage of power change | -0.10 (0.11) | -0.12 (0.12)
Statistical Analysis 1: Comparison: Personal Sound Amplification Products vs Control; Null hypothesis is that there was no difference in alpha power between PSAPs and Control. Data were analyzed using a linear mixed-effects (LME) model. The model included session (PSAPs, Control) and signal-to-noise ratio (SNR) as within-subject factors. Participants were included as a random factor; Test type: Superiority; p = 1.00, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Result of the pairwise comparisons for the SNR by Session interaction in the linear mixed model analysis

5. Primary Outcome: Alpha Power (8-12 Hz) During the Processing of the First Word in a Medium Noise Condition, With and Without PSAPs
Description: Alpha power (8-12 Hz) for a cluster of temporoparietal electrodes (T7, TP7, CP5), measured between 50 and 500 ms after the onset of the first word of the speech-in-noise task, under a medium noise condition (signal-to-noise ratio of 0 dB), with and without PSAPs. Alpha power was measured using temporal spectral evolution analysis with EEG. Values are baseline corrected with the pre-stimulus interval period (-500, 0 ms). Higher values indicate greater alpha power compared to the pre-stimulus interval period (i.e., event-related synchronization).
Time Frame: 1 hour
Population: One participant did not complete the EEG portion of the study. Two other participants were excluded due to noisy data.
Measure: Mean (Standard Deviation); unit: percentage of power change
Arm/Group | Personal Sound Amplification Products | Control
Number analyzed (Participants) | 25 | 25
percentage of power change | -0.09 (0.14) | -0.08 (0.15)
Statistical Analysis 1: Comparison: Personal Sound Amplification Products vs Control; [analysis description as in outcome 4, analysis 1]; Test type: Superiority — This p-value has been adjusted using the Bonferroni correction. The threshold for statistical significance was p = 0.05 (two-sided); p = 1.00, Mixed Models Analysis; Result of the pairwise comparisons for the SNR by Session interaction in the linear mixed model analysis

6. Primary Outcome: Alpha Power (8-12 Hz) During the Processing of the First Word in a High Noise Condition, With and Without PSAPs
Description: Alpha power (8-12 Hz) for a cluster of temporoparietal electrodes (T7, TP7, CP5), measured between 50 and 500 ms after the onset of the first word of the speech-in-noise task, under a high noise condition (signal-to-noise ratio of -3 dB), with and without PSAPs. Alpha power was measured using temporal spectral evolution analysis with EEG. Values are baseline corrected with the pre-stimulus interval period (-500, 0 ms). Higher values indicate greater alpha power compared to the pre-stimulus interval period (i.e., event-related synchronization).
Time Frame: 1 hour
Population: One participant did not complete the EEG portion of the study. Two other participants were excluded due to noisy data.
Measure: Mean (Standard Deviation); unit: percentage of power change
Arm/Group | Personal Sound Amplification Products | Control
Number analyzed (Participants) | 25 | 25
percentage of power change | -0.08 (0.11) | -0.01 (0.13)
Statistical Analysis 1: Comparison: Personal Sound Amplification Products vs Control; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.36, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Result of the pairwise comparisons for the SNR by Session interaction in the linear mixed model analysis

7. Secondary Outcome: Self-reported Measure of Listening Effort With and Without PSAPs
Description: Self-reported listening effort in the speech-in-noise task when using PSAPs and when using no device. Participants used a seven-point Likert scale to rate the listening effort required to complete the speech-in-noise task. The specific question was: "Using the scale in front of you, can you estimate how much effort it took you to understand the words in the presence of background noise? If you think that the amount of effort was between two numbers on the scale, it is fine for you to pick a fraction," with number 1 corresponding to "No effort" and number 7 corresponding to "Extreme effort." A high score indicates a greater listening effort.
Time Frame: 1 hour
Population: All participants who completed all study visits were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Personal Sound Amplification Products | Control
Number analyzed (Participants) | 28 | 28
score on a scale | 3.8 (1.1) | 4.2 (0.9)
Statistical Analysis 1: Comparison: Personal Sound Amplification Products vs Control; Null hypothesis is that there was no difference in listening effort between PSAPs and Control. The listening effort score was analyzed using a cumulative link mixed model. A logit link function with flexible thresholds was used. The model included Session (PSAPs, Control) and Block (1, 2, 3) as within-subject factors. Participants were included as a random factor; Test type: Superiority; p < 0.001, Cumulative link mixed model — The threshold for statistical significance was p = 0.05 (two-sided)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the first and second sessions, over a period of approximately one week.
Arm/Group | Personal Sound Amplification Products | Control
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/45/NCT05076045/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT05076045/ICF_001.pdf